CLINICAL TRIAL: NCT01165255
Title: Bupropion and Specific Cardiovascular Malformations
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114592; EPI40642 (Other: GSK); WEUSKOP4894 (Other: GSK)
Record Dates: First submitted 2010-07-01; First posted 2010-07-19 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Depressive Disorder; Pregnancy; Smoking Cessation
Keywords: congenital malformation; cardiovascular malformation; cardiovascular defect; antidepressants; pregnancy; first trimester; Bupropion; prevalence
MeSH Terms: conditions — Depressive Disorder; Smoking Cessation; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants born to women who were exposed to antidepressants: Women ages 12 through 49 (as of delivery date) who were dispensed an antidepressant between 01 January 1995 and 30 September 2004 from the original Bupropion study.
  Interventions: Drug: 3. Exposure to other antidepressants during the first trimester comparison cohort; Drug: 2. Exposure to bupropion outside the first trimester comparison cohort; Drug: 1. Exposure to bupropion during the first trimester

INTERVENTIONS:
Drug: 3. Exposure to other antidepressants during the first trimester comparison cohort — Exposure to other antidepressants during first trimester was classified in the original study using pharmacy claims submitted electronically to the Ingenix Research Database to indicate dispensing of other antidepressants. Infants were classified according to maternal exposure to other antidepressants during the first trimester. The first trimester was estimated as the earliest probable conception date through 91 days (13 weeks) following the latest probable conception date (based on delivery diagnosis codes). This study will refine the exposure classifications into infants born to women who were exposed only to one type of an antidepressant ("other antidepressant monotherapy"), or more than one type of an antidepressant ("other antidepressant mono or polytherapy") during the first trimester. A woman was considered exposed if there is at least one dispensing of another antidepressant during the first trimester of pregnancy.
Drug: 2. Exposure to bupropion outside the first trimester comparison cohort — Exposure to bupropion outside the first trimester was classified in the original study using pharmacy claims submitted electronically to the Ingenix Research Database to indicate a dispensing of bupropion. The comparison cohort ("bupropion exposure outside the first trimester") included women whose bupropion exposure occurred at least one month before the estimated date of conception and women whose bupropion exposure occurred after the first trimester, but before delivery. This study will refine the exposure classifications into infants born to women, who were exposed only to bupropion ("bupropion monotherapy"), or bupropion and another type of an antidepressant ("bupropion mono-or polytherapy") during the period outside the first trimester.
Drug: 1. Exposure to bupropion during the first trimester — Exposure to bupropion during the first trimester was classified in the original study using pharmacy claims submitted electronically to the Ingenix Research Database to indicate a dispensing of bupropion. Infants were classified according to maternal exposure to bupropion during the first trimester. The first trimester was estimated as the earliest probable conception date through 91 days (13 weeks) following the latest probable conception date (based on delivery diagnosis codes). This study will refine the exposure classifications into infants born to women, who were exposed only to bupropion ("bupropion monotherapy"), or bupropion and another type of an antidepressant ("bupropion mono-or polytherapy"). A woman was considered exposed in the first trimester if there was at least one dispensing of bupropion during the first trimester of pregnancy.

SUMMARY:
The study is an extension of earlier work based on a retrospective epidemiologic study of infants born to women who were exposed to bupropion in their estimated first trimester of pregnancy using data from a large US health plan affiliated with i3 Drug Safety (Clinical study ID WWE113694) (Cole JA, Oh KS, Chiang CC, Walker AM, Haight BR, Modell JG. Bupropion in pregnancy and the prevalence of congenital malformations Pharmacoepidemiology and Drug Safety, 2007; 16: 474-484). The cohorts developed for the earlier work consisted of all infants born to women exposed to bupropion during the estimated first trimester and outside the first trimester, and a random sample of infants born to women exposed to other antidepressants during the first trimester between 01 January 1995 and 30 September 2004. The objectives for this study include refining of both the original first trimester bupropion cohort and the original bupropion outside the first trimester cohort into mono-therapy and mono- or poly-therapy. Exposure to other antidepressants during the first trimester will also be refined into mono-therapy and mono- or poly-therapy. With input from pediatric cardiology expert, lists of specific cardiovascular malformations and malformation groupings will be created. The groupings will be created among the refined first trimester bupropion cohort as well as in two comparison cohorts of bupropion outside the first trimester and first trimester antidepressant use (mono-therapy and mono-or poly-therapy). The prevalence in each cohort will be calculated as the number of infants with a specific cardiovascular malformation divided by the number of live born infants. Prevalence will be reported per 1,000 infants. Confidence intervals will be calculated using Wilson's approximation to exact binomial intervals when the number of cases is five or greater and exact binomial intervals when the number of cases is fewer than five. The appropriateness of further calculations will be evaluated. Where numbers permit, adjusted odds ratios for specific cardiovascular groups/malformations will be calculated and if appropriate, stratified according to maternal dispensing of medications suspected to be teratogenic. The following comparisons, if numbers permit, will be performed: 1) bupropion first trimester mono-therapy cohort versus other antidepressant first trimester mono-therapy cohort; 2) bupropion first trimester mono- or poly-therapy cohort versus other antidepressant first trimester mono- or poly-therapy cohort; 3) bupropion first trimester mono-therapy cohort versus bupropion outside of first trimester mono-therapy cohort, and 4) bupropion first trimester mono- or poly-therapy cohort versus bupropion outside of first trimester mono- or poly-therapy cohort. Adjusted odds ratios will be calculated through a generalized estimated equations form of multivariate logistic regression to account for births associated with multiple infants. The same covariates identified in the original study will be included in this re-analysis. Covariates included: diagnoses of bipolar disorder and eclampsia within one year before delivery; dispensings of lithium, phenytoin, and fluconazole within one year before delivery through the end of the first trimester; and the number of physician visits within 10 to 12 months before delivery, maternal age, geographic region of the health plan, and infant gender. If generalized estimating equation form of the logistic regression model does not converge, adjusted odds ratios will be presented from a conventional multivariate logistic model. If the conventional multivariate logistic model does not converge, only the crude odds ratio will be presented.

DETAILED DESCRIPTION:
Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymised and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be the same as that used previously in the retrospective epidemiologic study of infants born to women who were exposed to bupropion in their estimated first trimester of pregnancy using data from a large US health plan affiliated with i3 Drug Safety.

* All deliveries occurring between 01 January 1995 and 30 September 2004 among women ages 12 to 49 who are members of UnitedHealthcare
* Eligible for prescription benefits
* Have one or more dispensings of an antidepressant during the study period
* Continuously enrolled for at least eighteen months prior to delivery
* Women were required to have one year of continuous health plan membership before their delivery date.
* Women were also included when the associated infant remained on the insurance plan.

Exclusion Criteria:

* Members who are employees of UnitedHealthcare are excluded from the Ingenix Research Database.

Ages: 12 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will be the same as that used previously in the retrospective epidemiologic study of infants born to women who were exposed to bupropion in their estimated first trimester of pregnancy using data from a large US health plan affiliated with i3 Drug Safety. 1,213 infants born to 1,140 women (1,142 pregnancies) were exposed to bupropion during the first trimester. The comparison groups consisted of 4,753 infants born to 4,617 women (4,649 pregnancies) exposed to other anti-depressants during the first trimester, and 1,049 infants born to 1,009 women (1,009 pregnancies) exposed to bupropion outside of the first trimester. All medical and prescription claims data along with dates of health plan enrollment for these women were included. The other antidepressant sample was frequency-matched to the bupropion cohort by year of birth, and was selected irrespective of exposure to specific antidepressants.
Sampling Method: Non-Probability Sample
Enrollment: 7005 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Frequencies and prevalence estimates of specific cardiovascular malformations and malformation groupings among live infants born to women exposed to bupropion or antidepressants | As performed previously, medical and prescription claims data was assembled and the outcomes of infants in the first 9 months of life were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline